CLINICAL TRIAL: NCT05637801
Title: A Randomized, Double-blind, Sham-controlled, Adaptive- Design Pivotal Study of Sensory Stimulation in Subjects With Alzheimer's Disease (Hope Study, CA-0011)
Brief Title: A Pivotal Study of Sensory Stimulation in Alzheimer's Disease (Hope Study, CA-0011)
Acronym: Hope
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cognito Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-0011
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Alzheimer Disease 1; Alzheimer Disease 2; Alzheimer Disease 3; Alzheimer Disease, Early Onset; Alzheimer Disease, Late Onset; Alzheimer Disease 9; Alzheimer Disease 4; Alzheimer Disease 7; Alzheimer Disease 17; Alzheimer's Dementia Late Onset; Alzheimer Disease 5; Alzheimer Disease 6; Alzheimer Disease 8; Alzheimer Disease 10; Alzheimer Disease 11; Alzheimer Disease 12; Alzheimer Disease 13; Alzheimer Disease 14; Alzheimer Disease 15; Alzheimer Disease 16; Alzheimer Disease 18; Alzheimer Disease 19; Dementia; Dementia Alzheimers; Dementia, Mild; Dementia of Alzheimer Type; Dementia Moderate; Dementia Senile; Mild Cognitive Impairment; Mild Dementia; MCI; Cognitive Impairment; Cognitive Decline; Cognitive Impairment, Mild
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Dementia; Gamma Stimulation; Cognito
MeSH Terms: conditions — Alzheimer Disease; Alzheimer disease type 1; Alzheimer disease type 2; Alzheimer disease, familial, type 3; Alzheimer Disease 9; Alzheimer disease type 4; Alzheimer Disease 7; Alzheimer Disease 5; Alzheimer Disease 6; Alzheimer Disease 8; Alzheimer Disease 10; Alzheimer Disease 11; Alzheimer Disease 12; Alzheimer Disease 13; Alzheimer Disease 14; Alzheimer Disease 15; Alzheimer Disease 16; Dementia; Lymphoma, Follicular; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Sham-controlled, Adaptive-Design Pivotal Study of Sensory Stimulation in Subjects with Alzheimer's Disease
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study; the investigator, the subject and study partner, and all other study personnel involved with subject assessments will remain blinded to the actual treatment assignment of the subjects. The Sponsor and their delegates involved in the study will be blinded to actual treatment assignment with the exception of technicians who are necessarily unblinded to assign and maintain the Investigational Devices and data analysis personnel as indicated in the Statistical Analysis Plan (SAP). Technicians and customer service agents who interact with subjects, their study partners and clinical sites will be specially trained to not reveal the study assignment (Active or Sham).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Treatment Group: Subjects are treated with the Active Sensory Stimulation System at home for 60 minutes daily for up to12 months.
  Interventions: Device: Sensory Stimulation System (GS120) - Active
- Control (Sham Comparator): Control Group: Subjects are treated with a Sham Sensory Stimulation System at home for 60 minutes daily for up to 12 months.
  Interventions: Device: Sensory Stimulation System (GS120) - Sham

INTERVENTIONS:
Device: Sensory Stimulation System (GS120) - Active — Sensory Stimulation System (GS120) - Active settings
  Arms: Active
Device: Sensory Stimulation System (GS120) - Sham — Sensory Stimulation System (GS120) - Sham settings
  Arms: Control

SUMMARY:
This is a randomized, double-blind, sham-controlled, adaptive-design pivotal study of sensory stimulation in subjects with mild to moderate Alzheimer's disease. Up to approximately 670 subjects will be randomized to 12 months of daily treatment with either Active or Sham Sensory Stimulation Systems. Efficacy will be measured using the Alzheimer's Disease Cooperative Study- Activities of Daily Living (ADCS-ADL) assessment and a combined statistical test (CST) of the ADCS-ADL and the Mini-Mental State Exam (MMSE).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, sham-controlled, adaptive design pivotal study.

The objective of the study will be to assess efficacy of gamma sensory stimulation (visual and audio) in slowing disease progression versus Sham for subjects with mild to moderate AD as measured functionally by the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) assessment and a combined statistical test (CST) for ADCS-ADL and the Mini-Mental State Exam (MMSE). Secondary objectives will include measures of cognition and neuroanatomical change.

Up to approximately six hundred and seventy (670) Mild to Moderate Alzheimer's disease subjects (MMSE 15-28) will be recruited at up to 70 clinical sites in the United States and randomized in a 1:1 ratio (Treatment: Control). In the Treatment Group, subjects will be treated with the Active Sensory Stimulation System once daily. In the Control Group, subjects are treated with a Sham Sensory Stimulation System once daily. Daily treatment is planned for up to 12 months.

Subjects will attend study visits for informed consent, screening and baseline, then at 3-Months, 6-Months, 9-Months (by phone), 12 Months and 13 Months (for safety follow-up).

Some clinical sites will be included in a substudy evaluating additional fluid biomarkers. Select participants enrolled at these sites will undergo a lumbar puncture to collect cerebrospinal fluid (CSF) at Baseline, 3 Months, and 12 Months.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women age 50-90
* Alzheimer's disease diagnosis with at least 6-month decline in cognitive function
* Non-childbearing potential or using adequate birth control
* Mini-Mental State Exam (MMSE) 15-28
* Available/consenting Study Partner
* Able to identify a Legally Authorized Representative (LAR)
* Stable chronic conditions at least 30 days
* Formal education of 8 or more years
* Adequate vision (Able to detect light) and hearing
* Mobility sufficient for compliance with testing procedures (ambulatory or aided-ambulatory, i.e. cane or walker)
* Amyloid or phosphorylated Tau positivity

Exclusion Criteria:

* Seizure disorder
* Hospitalization in previous 30 days
* Living in continuous care nursing home (assisted living permitted)
* Inability to have an MRI or significant abnormality on MRI screening
* Geriatric Depression Scale (GDS) >6
* Suicidality (current or previous 6 months)
* Serious neurological diseases affecting the Central Nervous System, including:

  1. other primary degenerative dementias (Lewy-body dementia, fronto-temporal dementia, Huntington's disease, Creutzfeldt-Jakob disease, Down syndrome, mixed dementia, etc),
  2. neurodegenerative conditions (Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis, etc),
  3. serious infection of the brain (meningitis/encephalitis), or
  4. history of multiple concussions.
* Metabolic or systemic diseases affecting the central nervous system (syphilis, B12 or folate deficiency, etc)
* Schizophrenia or bipolar disorder
* Heart disease, chronic liver, kidney, or respiratory disease, or uncontrolled diabetes or thyroid disease
* Cancer history within previous 2 years (except resolved non-melanoma skin or stable prostate)
* Nootropic drugs except stable acetylcholinesterase inhibitors
* Drug or Alcohol abuse in previous 12 months
* Previous exposure to Anti-amyloid-beta vaccines
* Past Exposure to Immunomodulators or passive immunotherapies for AD (ie, monoclonal antibodies)
* Exposure to BACE (β-Site amyloid precursor protein cleaving enzyme) inhibitors within the 6 months prior to consent
* Involved in a previous Cognito study or gamma therapy study
* Active treatment with Memantine (Namenda or Namzaric) within previous 30 days
* Life expectancy < 24 months

Participants involved in the Fluid Biomarker substudy also must not have contraindications to lumbar puncture.

For more information visit: https://www.hopestudyforad.com/

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Function as measured by the ADCS-ADL
Change from Baseline in Combined Statistical Test (CST) for Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) and Mini-Mental State Exam (MMSE) at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Function and Cognition as measured by CST for ADCS-ADL and MMSE

SECONDARY OUTCOMES:
Key Secondary: Change from Baseline in Mini-Mental State Exam (MMSE) at 12 Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Cognition as measured by MMSE
Change from Baseline in Whole brain volume at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Whole brain volume as measured by 3 Tesla (3T) Magnetic Resonance Imaging (MRI)
Change from Baseline in Hippocampal volume at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Hippocampal volume as measured by 3 Tesla (3T) Magnetic Resonance Imaging (MRI)
Change from Baseline in Clinical Dementia Rating- Sum of Boxes (CDR-SB) at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Global change in symptoms as measured by CDR

CONTACTS AND LOCATIONS:
Overall Officials: Robbert Zusterzeel, MD, PhD, MPH, Principal Investigator — Cognito Therapeutics
Locations (68):
- United States (68):
  - CCT Research - Gilbert Neurology Partners, Gilbert, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - CCT Research - Foothills Research Center, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Advanced Research Center, Inc, Anaheim, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neurology Center of North Orange County, Fullerton, California
  - Syrentis Clinical Research, Santa Ana, California
  - Office of Elizabeth Zarate-Rowell, MD, Seal Beach, California
  - Mile High Research Center, Denver, Colorado
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network- Aventura, Aventura, Florida
  - South Lake Pain Institute, Clermont, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Alphab Global Research, Jupiter, Florida
  - Charter Research - Lady Lake, Lady Lake, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Premier Clinical Research Institute Inc., Miami, Florida
  - Visionary Investigators Network- Miami, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Coastal Family Medicine - Orange Park, Orange Park, Florida
  - K2 Medical Research - Orlando, Orlando, Florida
  - Emerald Coast Neurology, Pensacola, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group - Sarasota, Sarasota, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Brain Matters Research, Stuart, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Charter Research - Winter Park, Winter Park, Florida
  - Emory Alzheimer's Disease Research Center, Atlanta, Georgia
  - NeuroStudies, Decatur, Georgia
  - Great Lakes Clinical Trials- Flourish Research- Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials- Flourish Research- Gurnee, Gurnee, Illinois
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Northern Light Acadia Hospital, Bangor, Maine
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Office of Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - Sisu BHR, LLC, Springfield, Massachusetts
  - QUEST Research Institute, Farmington, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - CCT Research - Papillion Research Center, Papillion, Nebraska
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - Alzheimer's Memory Center - AMC Research, Matthews, North Carolina
  - Insight Clinical Trials, LLC, Beachwood, Ohio
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Center for Cognitive Health - Portland, Portland, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Prisma Health Neurology, Columbia, South Carolina
  - Coastal Neurology, Port Royal, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - North Texas Clinical Trials, Fort Worth, Texas
  - UT Health San Antonio, Glenn Biggs Institute for Alzheimer's and Neurodegenerative Diseases, San Antonio, Texas
  - TRS Health, Stafford, Texas
  - Mercury Clinical Research, Sugarland, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - ReCogniton Health, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No